CLINICAL TRIAL: NCT04323176
Title: 2nd AC+: Leveraging Technology to Create Communities of Care Around Older People Living With HIV
Brief Title: 2nd AC+: New Village Model
Acronym: 2nd AC+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: The San Diego LGBT Community Center (Unknown)
Responsible Party: Principal Investigator, Maile Young Karris, Associate Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 182147; Age Positively (Other: Gilead Sciences)
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Aging; Hiv; Loneliness; Social Isolation
Keywords: HIV; Aging; Loneliness; social isolation; multi-morbidity; LGBT; community
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Social Isolation

STUDY DESIGN:
Intervention Model Description: Implementation of Village Model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Village Model (Experimental): Participate as a member of the Village using a website for 12 months.
  Interventions: Other: Village Model implementation

INTERVENTIONS:
Other: Village Model implementation — Participate in the Village Model using a website

SUMMARY:
This study evaluates implementation of the Village Model to support older people living with HIV.

DETAILED DESCRIPTION:
Understanding that older people living with HIV are facing uniques challenges as they age (lack of peer set due to extreme loss during the AIDS epidemic, ongoing HIV and age stigma, high rates of multi-morbidity) this study explores the acceptability and feasibility of implementing the Village Model in Central San Diego.

The Village Model started when several older members of Boston's Beacon Hill realized they were aging and may need more help as they aged to thrive in their own homes. The Village Model involves members of a community paying annual fees to support a village administrator that organizes regular socialization events and helps coordinate needs of individual members using the skill sets of other members within the community. From that first experience a few decades ago, today over 200 Villages exist across the country to enhance the ability of older adults to age in place.

However limitations of this model exists that may threaten the long term implementation and sustainability of the Village Model. Specifically the requirement to pay annual fees for an administrator, the lack of diversity (in age, race, sexuality etc), and difficulty in meeting member's needs in real-time.

This project proposes to pilot the Village Model in Central San Diego and will implement the following adaptions to address limitations. Members will not be required to pay annual fees but instead depend on a well-funded, long-established diverse organization (The San Diego LGBT Center) to serve as the administrator. This Village will allow participation of persons within the community at all ages, race, economic status. Lastly, the project proposes to pilot the acceptability of using a website to display and respond to community needs in real time.

To achieve this, the investigators will 1) perform questionnaires to understand the needs in the community by collecting needs assessments. 2) The investigators will explore the meaning of community and explore barriers and facilitators of Village Model implementation. 3) Lastly the investigators will pilot the Village model using a website.

ELIGIBILITY:
Inclusion Criteria:

* Lives in Central San Diego
* Consents to participate
* Willing to sign Village social contract
* No plans to move out of Central San Diego in the next year
* Speaks English

Exclusion Criteria:

* Severely cognitively impaired as indicated by < 10 on mini mental state examination
* History of a violent felony or fraud in the past 10 years
* Not willing to consent to participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Theoretical Framework Acceptability Scale | 12 months.
  A 7 question survey the investigators developed based on the Theoretical Framework of Acceptability. This likert scale includes answers on a 1-5 scale for each 7 questions. The range will be from 5-35 with higher scores indicating higher acceptability.

SECONDARY OUTCOMES:
Social Network Inventory | 1, 3, 6, and 12 months
  We will enumerate the social network of persons across four domains of support: emotional, material, social, and service. This will be done asking a series of questions about each persons named

OTHER OUTCOMES:
Engagement with the Village | 12 months
  Total count of times each study participant engaged in a Village request or event.
Engagement with the hyperlocal social app | 12 months
  Total count of times each study participant utilized the social app to request or provide a Village service

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The San Diego Lesbian Gay Bisexual Transgender Center, San Diego, California
  - University of California San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: Yes
On completion of the study, we will provide coded IDP to other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At study completion
Access Criteria: Please email study PI for requests. We will review to ensure work is not duplicative of ongoing analyses and that the intent of the work is not to exploit study participants.